CLINICAL TRIAL: NCT01246544
Title: Helsinki Declaration on Patient Safety
Acronym: Patient Safety
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Charite University, Berlin, Germany
Other Study IDs: Patient Safety
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Patient Safety
Keywords: Patient Safety; The Helsinki Declaration on Patient Safety in Anaesthesiology; Helsinki Declaration on Patient Safety; European Board of Anaesthesiology (EBA); European Society of Anaesthesiology (ESA)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data collection group: physicians: Online survey for physicians/members of the innovation alliance Berlin-Brandenburg (INABBRA)

SUMMARY:
In cooperation with INABBRA (Innovation Alliance Berlin-Brandenburg, Germany) the investigators would like to ask medical colleagues in the region to participate in an anonymous German online survey on patient safety.

The investigators want to investigate the implementation and establishment of measures on patient safety, that anaesthesiologists utilize to fulfill their obligations.

DETAILED DESCRIPTION:
The Declaration builds on earlier statements about safety and quality of care. It represents a shared European opinion of what currently is both worth doing and practical to improve patient safety in anaesthesiology in 2010. The Declaration recommends practical steps that all anaesthesiologists who are not already using them should include in their own practice. These are relatively straightforward and where they are currently being used have a track record of improving patient safety. All European anaesthesiology institutions are expected to support the World Health Organization(WHO) 'Safe Surgery Saves Lives' initiative including the "Safe Surgery Checklist". The Declaration was endorsed by European Board of Anaesthesiology (EBA) and the European Society of Anaesthesiology (ESA). It was officially launched at the Euroanaesthesia congress in Helsinki in June 2010 and was subsequently signed by several representatives of European anaesthesiology and different additional stakeholders (WHO, World Federation of Societies of Anaesthesiologists (WFSA), European Patients Federation (EPF)).

In cooperation with INABBRA (Innovation Alliance Berlin-Brandenburg, Germany) the investigators would like to ask medical colleagues in the region to participate in an anonymous German online survey on patient safety.

The investigators want to investigate the implementation and establishment of measures on patient safety, that anaesthesiologists utilize to fulfill their obligations under the perspective of the Declaration.

ELIGIBILITY:
Inclusion Criteria:

Members of the innovation alliance Berlin-Brandenburg (INABBRA)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Members of the innovation alliance Berlin-Brandenburg (INABBRA)
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Actual level on patient safety in Berlin-Brandenburg | 3 months
  Actual level on patient safety in Berlin-Brandenburg; comparing this to the recommendations of the Helsinki Declaration on Patient Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum/Campus Charité Mitte, Charité Universitätsmedizin, Berlin, State of Berlin, Germany